CLINICAL TRIAL: NCT00001489
Title: The Effect of Vigabatrin on Cerebral Blood Flow and Glucose Metabolism
Brief Title: Effect of Vigabatrin on Brain Blood Flow and Glucose Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950008; 95-N-0008
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Epilepsy; Epilepsy, Complex Partial
Keywords: Cerebral Metabolism; Complex Partial Seizures; Epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsy, Complex Partial; Seizures

SUMMARY:
This study is designed to test the effects of vigabatrin (gamma-vinyl-GABA) an experimental drug used for the treatment of epilepsy. The study will use positron emission tomography (PET scan) to detect areas of the brain receiving increased blood flow and using increased amounts of glucose. Increases in blood flow and glucose use are good indicators of brain activity.

Researchers are interested in determining the effects of Vigabatrin on brain blood flow and glucose use.

DETAILED DESCRIPTION:
This double-blind placebo-controlled parallel design protocol will investigate the effects of gamma-vinyl-GABA (vigabatrin--GVG) an experimental antiepileptic drug, on cerebral glucose metabolism (LCMRglc), blood flow (CBF), and seizure frequency, in patients with uncontrolled complex partial (CPS) and secondary generalized seizures (GTCS). Positron Emission Tomography (PET) will be used to measure CBF and LCMRglc.

ELIGIBILITY:
Localization-related epilepsy.

Uncontrolled seizures.

Ability to tolerate tegretol monotherapy.

No systemic illness requiring drug therapy.

No illness that might be made worse by vigabatrin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1994-10; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ben-Menachem E, Persson LI, Schechter PJ, Haegele KD, Huebert N, Hardenberg J, Dahlgren L, Mumford JP. The effect of different vigabatrin treatment regimens on CSF biochemistry and seizure control in epileptic patients. Br J Clin Pharmacol. 1989;27 Suppl 1(Suppl 1):79S-85S. doi: 10.1111/j.1365-2125.1989.tb03466.x. PMID 2474312
- [Background] Browne TR, Mattson RH, Penry JK, Smith DB, Treiman DM, Wilder BJ, Ben-Menachem E, Napoliello MJ, Sherry KM, Szabo GK. Vigabatrin for refractory complex partial seizures: multicenter single-blind study with long-term follow-up. Neurology. 1987 Feb;37(2):184-9. doi: 10.1212/wnl.37.2.184. PMID 3808298